CLINICAL TRIAL: NCT01692600
Title: Optical Coherence Tomography for Monitoring Late Oral Radiation Toxicity After Radiotherapy of Head and Neck Cancer Patients
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 12-0095-CE
Record Dates: First submitted 2012-08-30; First posted 2012-09-25 (Estimated); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Abnormalities, Radiation-Induced
Keywords: Late oral radiation toxicity; head and neck cancer patients; optical coherence tomography; subsurface imaging; mirometer-resolution imaging; vascular imaging; Doppler optical coherence tomography; speckle variance optical coherence tomography
MeSH Terms: conditions — Abnormalities, Radiation-Induced

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- healthy volunteers: Age-matched with the patient group, with no oral pathologies and comorbidities
- Late oral radiation toxicity patients: Head-and-neck cancer patients who had undergone radiation therapy and developed late radiation side ffects

SUMMARY:
Radiation therapy of the head and neck cancer patients causes late oral radiation complications such as xerostomia (dry mouth) or mucosal atrophy. Currently, methods such as hyperbaric oxygen are used to treat these complications; however, there are no quantifiable means of assessing the outcome of these methods. At present, subjective methods such as superficial examination of the oral cavity are used, yet complications are known to mostly start in the subsurface layers. In this feasibility study, we apply an imaging technique called optical coherence tomography (OCT) as a means of providing objective and quantifiable images of the subsurface micro-structural and micro-vascular changes of oral tissue. Depth-resolved, micrometer-resolution OCT images provide information on changes associated with late radiation complications.

DETAILED DESCRIPTION:
Patient imaging

At the imaging session, the patient will be asked to sit on the chair and put her/his chin on the chin-rest and the height of the chair will be adjusted accordingly. Before turning on the light source, the patient will be asked to wear the safety goggles and open her/his mouth while the probe is slowly moved inside the oral cavity. At this point, by looking at the superficial oral tissue, we will find regions in the oral cavity with superficial changes. When such regions are found, OCT images of these regions will be taken. Imaging of each location is expected to take about 3 to 4 minutes (including the time required to find the region of interest, acquisition of structural, Doppler and speckle variance images, and the time between each of these processes). After this, the patient can close her/his mouth and rest for couple of minutes. The same procedure will be performed on another site of complication. The 3-4 minute imaging procedure is repeated 3 to 5 times (depending on the patients' ability to keep the mouth open), after which the patient is dismissed and the sterile probe cover will be disposed. All the acquired data will be stored in a computer which is kept in a locked office. The data will be processed within the week after the imaging session so that structural, Doppler and speckle variance images of the imaged sites of complication can be compared.

During imaging, structural OCT real-time images are shown on the monitor to facilitate the task of finding the region of interest and keeping track of the patient's movements and move the probe accordingly. During the Doppler or speckle variance imaging (approximately 7 seconds each within the 3-4 minutes interval mentioned before), the patient is asked to keep as still as possible, in order to avoid any motion artifact in the OCT images.

Note that time frame for this study is 1 day, since subjects are only imaged once with no follow-up assessments.

Imaging healthy volunteers

The imaging session of the volunteers takes between 30 to 60 minutes. The imaging procedure of these healthy volunteers is very similar to that explained for the patients; however, all the acquired OCT images of this group would be of healthy oral tissue.

Note that time frame for this study is 1 day, since the volunteers are only imaged once with no follow-up assessments.

**Important note: The aim of this study is to compare the images from patients with those of healthy volunteers and show that there are specific changes in the structural and vascular features of the patients (due to radiation toxicity) when compared to the volunteers. So, the comparison is done between the two cohorts of the study.

Data analysis

For the healthy volunteers, the gathered OCT data will be processed to form structural, Doppler and speckle variance images of healthy oral tissue to serve as a reference. The same procedure will be performed on late oral radiation toxicity patients to reconstruct structural, Doppler and speckle variance images of the site of oral complications. Then, the images of healthy volunteers and patients will be compared in terms of the layer thickness, the back-reflection properties of each layer, and the size and profile of blood flow of the microvasculature. In order to compare these two sets of images quantitatively, certain metrics will be defined based on the images of the healthy volunteers. All these quantitative comparisons of healthy oral tissue and tissue with radiation complication will be used to form an OCT atlas of oral radiation toxicity. Moreover, white-light images of the regions of OCT study will be taken in order to serve as a reference for the superficial complications caused by radiation.

ELIGIBILITY:
for the patients:

1. Must have undergone radiation therapy of the head and neck site
2. Must have developed some form of late oral radiation toxicity
3. Attending the radiation late effects clinic at Princess Margaret Cancer Center, Toronto, Canada

For the healthy volunteers:

1- Generally healthy

Exclusion criteria for the patients:

1. Unable to keep the mouth open for more than 3 minutes
2. Unable to open the mouth more than 2cm (to admit the OCT probe)
3. Having loose teeth

for the healthy volunteers:

1. Having an oral infection or disease
2. Unable to keep the mouth open continuously for 5 minutes
3. Unable to open the mouth more than 2cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population are selected from the patients who have received radiation as a treatment for head and neck cancer and have developed late radiation toxicity in their oral tissue. This population is selected among the patients who can open their mouth more than 2 centimeters (so that the imaging probe can be inserted into their oral cavity)
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Comparison between the oral layer structure of radiation toxicity patients and healthy volunteers as shown in the OCT structural images | at the imaging time point [comparison between cohorts]
  Structural OCT images of the oral tissue of the late radiation toxicity patients will be taken and will be processed to highlight any differences between them and the healthy human oral tissue. An example of the expected differences (in the patients compared to healthy volunteers) is total loss of basal layer and thus loss of differentiation between epithelium and lamina propria in the patients.

SECONDARY OUTCOMES:
Comparison between vascular structure and blood flow properties in the vascular OCT images of radiation toxicity patients and healthy volunteers as shown in the OCT vascular images | At the imaging time point [comparison between cohorts]
  Doppler OCT and speckle variance OCT images will be taken to reveal information on the blood flow and vascular structure, respectively. These images will be processed and information about the blood flow, size of the vasculature, and vessel density of the radiation toxicity patients will be extracted and the average values will be compared to those of healthy human volunteer cases

CONTACTS AND LOCATIONS:
Overall Officials: Alex I Vitkin, PhD, Principal Investigator — University of Toronto/UHNToronto
Locations (1):
- Princess Margaret Hospital/UHNTorotno, Toronto, Ontario, Canada

REFERENCES:
- [Background] Davoudi B, Lindenmaier A, Standish BA, Allo G, Bizheva K, Vitkin A. Noninvasive in vivo structural and vascular imaging of human oral tissues with spectral domain optical coherence tomography. Biomed Opt Express. 2012 May 1;3(5):826-39. doi: 10.1364/BOE.3.000826. Epub 2012 Apr 2. PMID 22567578
- [Result] Davoudi B, Morrison M, Bizheva K, Yang VX, Dinniwell R, Levin W, Vitkin IA. Optical coherence tomography platform for microvascular imaging and quantification: initial experience in late oral radiation toxicity patients. J Biomed Opt. 2013 Jul;18(7):76008. doi: 10.1117/1.JBO.18.7.076008. PMID 23843086
- [Result] Davoudi B, Bizheva K, Wong A, Dinniwell R, Levin L and Vitkin A. Correlating optical coherence tomography images with dose distribution in late oral radiation toxicity patients. Photonics and Lasers in Medicine 3(4): 311-321, 2014